CLINICAL TRIAL: NCT03774017
Title: Study on Benefits and Risks of Hybrid Operation in the Treatment of Complex Brain Arteriovenous Malformations
Brief Title: Research on Hybrid Operation Technique in the Treatment of Complex Brain Arteriovenous Malformations
Acronym: HOTAVM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Shuo Wang, Director of Neurosurgery Department, Ministry of Science and Technology of the People´s Republic of China
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BJTTH-007; 2016YFC1301801 (Other Grant/Funding Number: National Key Technologies R&D Program of China)
Record Dates: First submitted 2018-12-11; First posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Cerebrovascular Disease; Arteriovenous Malformations; Complex; Primary
Keywords: brain arteriovenous malformations; one-staged hybrid operation
MeSH Terms: conditions — Cerebrovascular Disorders; Arteriovenous Malformations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional microsurgery group (Other): Patients receive only traditional microsurgical operations in traditional operating theaters or the one-staged hybrid operation theater. No endovascular intervention technique or intraoperative digital subtraction angiography(DSA) will be performed. The DSA will be performed in 3 days after the operation.
  Interventions: Procedure: Traditional microsurgical operation
- Hybrid operation group (Experimental): Patients receive microsurgical operation under the assistance of intraoperative DSA, endovascular embolization and/or balloon occlusion in the one-staged hybrid operating theater.
  Interventions: Procedure: one-staged hybrid operation

INTERVENTIONS:
Procedure: one-staged hybrid operation — An integrated procedure that consists of microsurgery, intraoperative DSA, endovascular intervention techniques and other assistance tools. All the procedures are performed in a one-staged operation without any intermission or any transfer of patients.
  Arms: Hybrid operation group
Procedure: Traditional microsurgical operation — The classical mode of operations in neurosurgery. The operation is performed with neurosurgical instruments and microscope. Some of assisting tools can be used in the operation, such as neuro-navigation, Doppler probe, neural electrophysiological monitoring and so on. But neither the intraoperative DSA nor endovascular intervention techniques is used in the operation
  Arms: Traditional microsurgery group

SUMMARY:
Complex brain arteriovenous malformations (bAVMs) in ≥3 Spetzler-Martin grades have long been challenges among cerebrovascular diseases. None of the traditional methods, such as microsurgical operation, endovascular intervention, or stereotactic radiotherapy, can completely eliminate complex bAVMs without a risk of neural function deterioration. The multistaged hybrid operation solved part of the challenge but remained risky in the installment procedures and intervals. The one-staged hybrid operation was applied in the surgical treatment of cerebrovascular diseases and proved to be a potentially safe and effective method for curing complex bAVMs. However, lacking the support of high-level evidence, its advantages remain unclear. This study was proposed to validate the benefits and risks of one-staged hybrid operation in the treatment of complex bAVMs, as well as its indications, key technologies, and workflows.

DETAILED DESCRIPTION:
The study is being conducted from Jan 2016 to Dec 2020 with 20 cooperation units. It consists of 2 sets. The registry set is designed as a prospective real-world registry. The trial set is designed as a prospective pragmatic clinical trial, specifically for the patients with perforating arterial feeders. The two sets share a common grouping: the traditional operation group and the one-staged hybrid operation group. The assignment is based on the clinical condition in the registry set and is randomized in the trial set. End points will be evaluated at scheduled time points. The safety and efficiency of one-staged hybrid operation in treating complex bAVMs will be validated.

ELIGIBILITY:
Inclusion Criteria:

1. patients of all ages;
2. diagnosed with arteriovenous malformations (AVMs) in brain parenchyma (including cerebrum and cerebellum) by DSA, with/without dura arteriovenous fistula;
3. with any operative indications as follows: (1) with stable hematoma or history of hemorrhage due to bAVMs, and allowed selective operation; (2) with recurrent epilepsy seizure, having failed treatment with antiepileptic drugs (AEDs); (3) with induced deterioration of neurological functions;
4. with Spetzler-Martin Grades from I to IV;
5. who provide informed consent.

Exclusion Criteria:

1. >70 years old with no significant hemorrhagic risk of bAVMs;
2. with Spetzler-Martin Grade ≥V;
3. accompanied by severe chronic disease, organ dysfunction, or malignant tumor that cannot tolerate the operation;
4. allergic to iodinated contrast agent;
5. unable to give informed consent.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
neural function deterioration | 3 months after operation
  Increasing of mRS and mRS>2

SECONDARY OUTCOMES:
neural function deterioration in 6 months | 6 months after operation
  Increasing of mRS and mRS>2
neural function deterioration in 12 months | 12 months after operation
  Increasing of mRS and mRS>2
postoperative mortality | 7 days after operation
  the fatality due to operation
operation-related complications | 7 days after operation
  any complications that occur within 7 days from the date of operation, including intracranial hemorrhage or infarction, infection of the central nervous system, infection of the respiratory system, cranial nerve deficits, and other symptomatic complications
postoperative bAVMs residue | 7 days after operation
  the bAVMs residue revealed by postoperative DSA or computed tomographic angiography
3 months bAVMs residue | 3 months after operation
  the bAVMs residue revealed by postoperative DSA or computed tomographic angiography
6 months bAVMs residue | 6 months after operation
  the bAVMs residue revealed by postoperative DSA or computed tomographic angiography
12 months bAVMs residue | 12 months after operation
  the bAVMs residue revealed by postoperative DSA or computed tomographic angiography

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Wang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (7):
- China (7):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital Capital Medical University, Beijing, Beijing Municipality
  - General Hospital of Rocket Army, Beijing, Beijing Municipality
  - Qilu Hospital, Shandong University, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang M, Qiu H, Cao Y, Wang S, Zhao J. One-staged in situ embolization combined with surgical resection for eloquence protection of AVM: technical note. Neurosurg Rev. 2019 Sep;42(3):783-790. doi: 10.1007/s10143-019-01137-w. Epub 2019 Jul 30. PMID 31359304
- [Derived] Wang M, Jiao Y, Cao Y, Wang S, Zhao J. Surgical management of complex brain arteriovenous malformations with hybrid operating technique: study protocol of a prospective registry and a pragmatic clinical trial. BMC Neurol. 2019 Apr 30;19(1):75. doi: 10.1186/s12883-019-1289-3. PMID 31039755